CLINICAL TRIAL: NCT04451720
Title: A Phase 3, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Risankizumab in Adult Japanese Subjects With Moderate to Severe Palmoplantar Pustulosis
Brief Title: Study of Subcutaneous Risankizumab Injection to Assess Change in Palmoplantar Pustulosis Area and Severity Index [PPPASI] in Adult Japanese Participants With Palmoplantar Pustulosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M19-135
Record Dates: First submitted 2020-06-29; First posted 2020-06-30 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Palmoplantar Pustulosis (PPP)
Keywords: Palmoplantar Pustulosis (PPP); Risankizumab; SKYRIZI
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risankizumab (Experimental): In Period A, participants will receive risankizumab dose A at Weeks 0 and 4. In Period B, participants will receive risankizumab dose A at Weeks 16, 28, 40 and 52, and also placebo at Weeks 20, 32, 44 and 56.
  Interventions: Drug: Risankizumab; Drug: Placebo
- Placebo (Experimental): In Period A, participants will receive placebo at Weeks 0 and 4. In period B, participants will receive risankizumab dose A at Weeks 16, 20,32,44 and 56. and also placebo at Weeks 28,40 and 52.
  Interventions: Drug: Risankizumab; Drug: Placebo

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous (SC) injection
  Other Names: SKYRIZI; ABBV-066
Drug: Placebo — Subcutaneous (SC) injection

SUMMARY:
Palmoplantar pustulosis is a chronic inflammatory skin disease that causes repeated on and off symptoms like erythema (reddening, irritation), vesicle (swelling, cyst), pustules, scale, and crusts in palms and soles. This study evaluates how well risankizumab works compared to placebo (no medicine) to treat palmoplantar pustulosis. Study will assess change in Palmoplantar Pustulosis Area and Severity Index [PPPASI].

Risankizumab is an investigational drug being developed for the treatment of palmoplantar pustulosis. This study is "double-blinded", which means that neither the trial participants nor the study doctors will know who will be given study drug and who will receive placebo (no medicine). Participants are randomly put into 1 of 2 groups, called treatment arms to receive risankizumab or placebo in period A. In period B, each group receives both risankizumab and placebo at different time intervals. Around 116 adult participants with palmoplantar pustulosis will be enrolled in approximately 39 sites across Japan.

Participants will receive subcutaneous (SC) injections of risankizumab or placebo at Week 0 and Week 4 (Period A). Beginning Week 16 (Period B), both the groups will receive risankizumab and placebo at different intervals. Total treatment duration is 56 weeks.

There may be a higher burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Stable moderate to severe Palmoplantar Pustulosis (PPP) with a Palmoplantar Pustulosis Area and Severity Index (PPPASI) total score of >= 12 at the Screening and Baseline Visits.
* Moderate or severe pustules/vesicles on at least one palm or sole (>= 2 PPPASI severity score) at the Screening and Baseline Visits.
* Experienced inadequate response (or intolerant) to treatment with topical corticosteroids and/or vitamin D3 derivative preparations and/or phototherapy and/or systemic etretinate.

Exclusion Criteria:

- History of active skin disease other than PPP which could interfere with the assessment of PPP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Palmoplantar Pustulosis Area and Severity Index (PPPASI) Total Score | Baseline (Week 0) through Week 16
  The Palmoplantar Pustulosis Area and Severity Index (PPPASI) assesses the severity of palmoplantar pustulosis lesions and their response to therapy. In the PPPASI system, the palms and soles are divided into 4 regions: the right palm, left palm, right sole, left sole which account for 20%, 20%, 30%, and 30%, respectively, of the total surface area of the palms and soles. Each of these areas are assessed separately for erythema, pustules/vesicle and desquamation/scale, which are each rated on a scale of 0 to 4. The PPPASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.

SECONDARY OUTCOMES:
Percentage of Participants Achieving at least 50% Improvement in PPPASI (PPPASI-50) | Baseline (Week 0) through Week 16
  The Palmoplantar Pustulosis Area and Severity Index (PPPASI) assesses the severity of palmoplantar pustulosis lesions and their response to therapy. In the PPPASI system, the palms and soles are divided into 4 regions: the right palm, left palm, right sole, left sole which account for 20%, 20%, 30%, and 30%, respectively, of the total surface area of the palms and soles. Each of these areas are assessed separately for erythema, pustules/vesicle and desquamation/scale, which are each rated on a scale of 0 to 4. The PPPASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving at least 75% Improvement in PPPASI (PPPASI-75) | Baseline (Week 0) through Week 16
  The Palmoplantar Pustulosis Area and Severity Index (PPPASI) assesses the severity of palmoplantar pustulosis lesions and their response to therapy. In the PPPASI system, the palms and soles are divided into 4 regions: the right palm, left palm, right sole, left sole which account for 20%, 20%, 30%, and 30%, respectively, of the total surface area of the palms and soles. Each of these areas are assessed separately for erythema, pustules/vesicle and desquamation/scale, which are each rated on a scale of 0 to 4. The PPPASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (39):
- Japan (39):
  - Ichinomiya Municipal Hospital /ID# 222581, Ichinomiya-shi, Aichi-ken
  - Chukyo Hospital /ID# 218894, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 221258, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 221285, Toyoake-shi, Aichi-ken
  - Toho University Sakura Medical Center /ID# 220858, Sakura-shi, Chiba
  - Ehime University Hospital /ID# 221260, Toon-shi, Ehime
  - Kurume University Hospital /ID# 222751, Kurume-shi, Fukuoka
  - Fukushima Medical University Hospital /ID# 221639, Fukushima, Fukushima
  - Gifu University Hospital /ID# 219109, Gifu, Gifu
  - Ogaki Municipal Hospital /ID# 220801, Ogaki-shi, Gifu
  - Takagi Dermatology Clinic /ID# 220896, Obihiro-shi, Hokkaido
  - Bito Dermatology Clinic /ID# 222750, Kobe, Hyōgo
  - Meiwa Hospital /ID# 221633, Nishinomiya-shi, Hyōgo
  - Ibaraki Prefectural Central Hospital /ID# 222712, Kasama-shi, Ibaraki
  - Mito Kyodo General Hospital /ID# 220799, Mito, Ibaraki
  - Takamatsu Red Cross Hospital /ID# 221344, Takamatsu, Kagawa-ken
  - Tokai University Hospital /ID# 220945, Isehara-shi, Kanagawa
  - National Hospital Organization Sagamihara National Hospital /ID# 219082, Sagamihara-shi, Kanagawa
  - Yokohama City University Hospital /ID# 220860, Yokohama, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine /ID# 221376, Kyoto, Kyoto
  - National Hospital Organization Kyoto Medical Center /ID# 221772, Kyoto, Kyoto
  - Mie University Hospital /ID# 221570, Tsu, Mie-ken
  - Tohoku University Hospital /ID# 219017, Sendai, Miyagi
  - Shinshu University Hospital /ID# 221343, Matsumoto-shi, Nagano
  - Nagasaki University Hospital /ID# 221141, Nagasaki, Nagasaki
  - Nagaoka Red Cross Hospital /ID# 221375, Nagaoka-shi, Niigata
  - Isonokami dermatological clinic /ID# 219023, Daito-shi, Osaka
  - Kansai Medical University Kori Hospital /ID# 223096, Neyagawa, Osaka
  - Osaka Metropolitan University Hospital /ID# 222012, Osaka, Osaka
  - Kindai University Hospital /ID# 219022, Osakasayama-shi, Osaka
  - Kume Clinic /ID# 220869, Sakai-shi, Osaka
  - Dokkyo Medical University Saitama Medical Center /ID# 222526, Koshigaya-shi, Saitama
  - Shizuoka Saiseikai Genaral Hospital /ID# 222427, Shizuoka, Shizuoka
  - Dokkyo Medical University Hospital /ID# 221210, Shimotsuga-gun, Tochigi
  - St.Luke's International Hospital /ID# 219019, Chuo-ku, Tokyo
  - Teikyo University Hospital /ID# 221089, Itabashi-ku, Tokyo
  - The Jikei University Hospital /ID# 218822, Minato-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 218893, Shinjuku-ku, Tokyo
  - Seibo Hospital /ID# 221691, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/